CLINICAL TRIAL: NCT04872166
Title: An Open Label, Escalating Multiple Dose Study to Evaluate the Safety, Toxicity, and Pharmacokinetics of BTX A51 Alone and in Combination With Fulvestrant in Subjects With Advanced Solid Tumors and Estrogen Receptor Positive, Human Epidermal Growth Factor Receptor 2 Negative Metastatic Breast Cancer
Brief Title: A Study of BTX-A51 in People With Advanced Solid Tumor and Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Edgewood Oncology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BTX-A51-002
Record Dates: First submitted 2021-04-22; First posted 2021-05-04 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Advanced Solid Tumor; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- BTX-A51 Dose Cohort 1 (Experimental): Starting dose (SD) of BTX-A51 administered orally 5 times per week in a 28-day cycle
  Interventions: Drug: BTX-A51
- BTX-A51 Dose Cohort 2 (Experimental): Up to 2-times the SD of BTX-A51 administered orally 5 times per week in a 28-day cycle
  Interventions: Drug: BTX-A51
- BTX-A51 Dose Cohort 3 (Experimental): Up to 3.5-times the SD of BTX-A51 administered orally 5 times per week in a 28-day cycle
  Interventions: Drug: BTX-A51
- BTX-A51 Dose Cohort 4 (Experimental): Up to 5-times the SD of BTX-A51 administered orally 5 times per week in a 28-day cycle
  Interventions: Drug: BTX-A51
- BTX-A51 Dose Cohort 5 (Experimental): Up to 7-times the SD of BTX-A51 administered orally 5 times per week in a 28-day cycle
  Interventions: Drug: BTX-A51
- BTX-A51 Dose Cohort 6 (Experimental): Up to 10-times the SD of BTX-A51 administered orally 5 times per week in a 28-day cycle
  Interventions: Drug: BTX-A51
- BTX-A51 in Combination with Fulvestrant Cohort 1 (Experimental): Starting dose (SD) of BTX-A51 administered orally 3 times per week in a 28-day cycle; fulvestrant administered as a 500-mg intramuscular injection on days 1 and 15 of cycle 1 and on day 1 of subsequent 28-day cycles.
  Interventions: Drug: BTX-A51
- BTX-A51 in Combination with Fulvestrant Cohort 2 (Experimental): Up to 2-times the SD of BTX-A51 administered orally 3 times per week in a 28-day cycle; fulvestrant administered as a 500-mg intramuscular injection on days 1 and 15 of cycle 1 and on day 1 of subsequent 28-day cycles.
  Interventions: Drug: BTX-A51

INTERVENTIONS:
Drug: BTX-A51 — One 28 day cycle of treatment will consist of 4 weeks of treatment with a weekly dosing schedule of up to 5 days per weekf.

SUMMARY:
This is a multicenter, open label, nonrandomized, sequential dose escalation/dose ranging, multiple dose study designed to evaluate the safety, toxicity, and PK as well as preliminary efficacy of BTX-A51 alone and in combination with fulvestrant in subjects with advanced solid tumors. The study will be done in three phases, described below.

Phase 1a (Dose Escalation Phase):

The Phase 1a portion is designed to determine the dose limiting toxicities (DLTs), maximum tolerated dose (MTD), and recommended Phase 2 dose (RP2D) of orally administered BTX-A51. BTX-A51 will be administered once daily on a weekly schedule of 5 days on/2 days off. Dose escalation will proceed according to a modified 3+3 design. Each cycle will consist of 28 days (4 weeks), and the DLT observation period will be the first cycle (i.e., 28 days after initiation of dosing). A DLT may be observed in no more than 0 out of 3 or 1 out of 6 subjects who have completed the DLT observation period before the next cohort initiates accrual. Barring DLT, sequential dose escalation of BTX-A51 is planned with up to a total of 6 dose levels; on the basis of these an MTD will be identified. The MTD is defined as the highest dose level with a subject incidence of DLTs of 0 or 1 out of 6 during the first 28 days of study drug dosing. A minimum of 6 subjects needs to be treated at a dose level before this dose level can be deemed as the MTD.

Phase 1b (Monotherapy Dose Ranging Phase):

Dose expansion may begin when the RP2D has been determined. Up to 40 additional subjects at each of the 2 dose levels will be enrolled to evaluate safety and preliminary efficacy of BTX-A51 in subjects with estrogen receptor positive (ER+), human epidermal growth factor receptor 2 negative (HER2-), GATA3 mutant (mt) and wild-type (wt) metastatic breast cancer (mBC). Dosing in this phase of the study consists of the first cycle of therapy (i.e., 28 days).

Phase 1c (Combination Safety Phase):

The Phase 1c portion will evaluate the safety and tolerability of orally administered BTX-A51 at two dose levels combined with fulvestrant. The first combo cohort may be initiated after DEC review of the 6 subject lead-in phase of the high dose monotherapy cohort in Phase 1b. Dose escalation will proceed according to a 3+3 design. Each cycle will consist of 28 days (4 weeks), and the DLT observation period will be the first cycle (i.e., 28 days after initiation of dosing).

ELIGIBILITY:
Inclusion Criteria:

* Demonstration of understanding and voluntarily signing of an informed consent form
* Age ≥ 18 years
* Histologically or cytologically documented, incurable or metastatic solid tumor that is refractory to or intolerant of all standard therapy or for which no standard therapy is available
* Phase 1b and 1c only: Histologically confirmed diagnosis of ER+, HER2- mBC not amenable to resection or radiation therapy with curative intent.
* Measurable disease per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1).
* Adequate organ function
* Females of childbearing age must not be pregnant at time of Screening/beginning of treatment and agree to either abstain from sexual intercourse or use highly effective methods of contraception (for up to 3 months after last dose of study drug)
* Males sexually active with a woman of childbearing age must agree to use barrier method of birth control during and after the study (up to 3 months after last dose of study drug)

Exclusion Criteria:

* Life expectancy <3 months, as determined by the Investigator.
* Treatment with any local or systemic antineoplastic therapy (including chemotherapy, hormonal therapy, or radiation) within 3 weeks prior to first dose of BTX-A51
* Chronic use of corticosteroids in excess of 10 mg daily of prednisone or equivalent within 4 weeks prior to first dose of BTX-A51
* Major trauma or major surgery within 4 weeks prior to first dose of BTX-A51.
* Adverse events from prior anti-cancer therapy that have not resolved to Grade ≤1 except for alopecia or Grade ≤2 immunotherapy-related thyroid toxicity.
* History of, or known, central nervous system (CNS) disease involvement, or prior history of NCI CTCAE Grade ≥3 drug-related CNS toxicity.
* Clinically significant cardiac disease
* Active uncontrolled systemic fungal, bacterial, mycobacterial, or viral infection
* Known positive test result for human immunodeficiency virus (HIV) or acquired immune deficiency syndrome (AIDS)
* Active hepatitis C virus (HCV) or hepatitis B virus (HBV)
* Second primary malignancy that has not been in remission for greater than 3 years
* Any serious underlying medical (e.g., pulmonary, renal, hepatic, gastrointestinal, or neurological) or psychiatric condition (e.g., alcohol or drug abuse, dementia or altered mental status) or any issue that would limit compliance with study requirements
* Pregnant, lactating, or breastfeeding.
* Participation or plans to participate in another interventional clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2021-06-07 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events after BTX-A51 administration alone and in combination with fulvestrant | From first dose of BTX-A51 through 30 days after the last BTX-A51 alone and in combination with fulvestrant treatment (subjects will be offered continued access to study BTX-A51 until disease progression or unacceptable toxicity)
  To examine the incidence of clinical and laboratory adverse events after multiple doses of BTX-A51 alone and in combination with fulvestrant.
Defining the maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D) of BTX-A51alone and in combination with fulvestrant | At the end of Cycle 1 (each cycle is 28 days)
  To assess number of patients experiencing dose-limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years after the last treatment or upon death.
  To evaluate the objective response rate (ORR) as determined by the specific disease response criteria
Duration of response (DoR) | Up to 2 years after the last treatment or upon death.
  To evaluate the duration of response (DoR), defined as time from the date of first documentation of response to the date of the first documentation of progressive disease (PD), or death due to any cause
Progression free survival (PFS) | Up to 2 years after the last treatment or upon death.
  To examine the the progression free survival (PFS), defined as time from the date of first dose of study treatment to the first date of documentation of PD, or death due to any cause
Overall survival (OS) | Up to 2 years after the last treatment or upon death.
  To examine the overall survival (OS), defined as time from the date of first dose of study treatment to death due to any cause
Peak Plasma Concentration of BTX-A51 | PK samples are collected at pre-dose and post-dose at 1, 2, 3, 5, 8, and 24 hours on Days 1 and 5 of Cycle 1 (each cycle is 28 days).
  To evaluate the maximum observed concentration (Cmax) after single and repeated oral, once daily doses of BTX-A51
Area under the plasma concentration of BTX-A51 | PK samples are collected at pre-dose and post-dose at 1, 2, 3, 5, 8, and 24 hours on Days 1 and 5 of Cycle 1 (each cycle is 28 days).
  To evaluate the area under the curve (AUC) plasma-concentration after single and repeated oral, once daily doses of BTX-A51
Half-life of BTX-A51 | PK samples are collected at pre-dose and post-dose at 1, 2, 3, 5, 8, and 24 hours on Days 1 and 5 of Cycle 1 (each cycle is 28 days).
  To evaluate the half-life of BTX-A51 after single and repeated oral, once daily doses of BTX-A51

CONTACTS AND LOCATIONS:
Overall Officials: Zung Thai, MD, Study Director — Edgewood Oncology Inc.
Locations (6):
- United States (6):
  - Florida Cancer Specialists, Lake Mary, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - The Linder Research Center at The Christ Hospital, Cincinnati, Ohio
  - SCRI Oncology Partners, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Ball BJ, Xiao W, Borthakur G, Nguyen LXT, Valerio M, Venkatachalam A, Marcucci G, Stein AS, Thai DL, Cook DN, Chan K, Persaud S, Levine RL, Abdel-Wahab O, Ben-Neriah Y, Stein EM. Phase I first-in-human dose escalation study of the oral casein kinase 1alpha and cyclin dependent kinase 7/9 inhibitor BTX A51 in advanced MDS and AML. J Hematol Oncol. 2025 Jul 15;18(1):73. doi: 10.1186/s13045-025-01724-z. PMID 40665325